CLINICAL TRIAL: NCT01836354
Title: Discharge Educational Strategies for Reduction of Vascular Events
Acronym: DESERVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Columbia University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-00718
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Intracerebral Infarcts; Ischemic Stroke; Hemorrhagic Strokes; TIA's
Keywords: stroke; interactive educational intervention; acute ischemic stroke; transient ischemic attack
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DESERVE education (Active Comparator): Intervention group will receive education on stroke preparedness plus risk factor reduction education, and help accessing follow up care with health workers.
  Interventions: Behavioral: DESERVE education
- Usual Care (No Intervention): The usual care group will only receive written preparedness education, which is the standard care for the hospital.

INTERVENTIONS:
Behavioral: DESERVE education — Those patients assigned to education will receive stroke comprehensive intervention which focuses on three main areas, Risk perception, Medication Adherence, and Patient-Physician Communication. We will test whether phone calls and visits with a health worker after discharge, videos and a workbook are linked to better control of blood pressure and other risk factors
  Arms: DESERVE education

SUMMARY:
DESERVE is a discharge education study using health workers to enroll and randomly assign 800 subjects diagnosed with TIA, or mild stroke to either risk factor education or usual care. Those patients assigned to education will receive stroke preparedness education plus risk factor reduction education, and help accessing follow up care with health workers. Those patients assigned to usual care will receive written stroke preparedness education. This protocol will evaluate the effectiveness of this intervention to reduce blood pressure, and individual stroke risk factors and future stroke risk.

DETAILED DESCRIPTION:
Stroke and its risk factors disproportionately affect minority populations, and secondary stroke prevention programs have had relatively little success. TIA and mild stroke patients with few after-affects also stay in the hospital for a shorter period of time, and leave without enough information about their risk for another stroke. Additionally, mild stroke and TIA patients often do not follow-up with neurologists after they leave the hospital. DESERVE is a discharge education study using health workers to enroll and randomly assign 800 subjects from MSSM, MSSM Queens and CUMC diagnosed with Transient Ischemic attack (TIA ), mild Ischemic stroke (IS) or mild Intracerebral Hemorrhage (ICH) to either risk factor education or usual care. Those patients assigned to education will receive education on stroke preparedness education plus risk factor reduction education, and help accessing follow up care with health workers. This education includes a power point presentation and a patient-paced workbook and video on Risk perception, Medication Adherence, and Patient-Physician Communication. To target the most appropriate mild IS/ICH and TIA survivors for participation in this proposal, we will focus on survivors with mild stroke and TIA, excluding those whose stroke deficits are severe enough to warrant discharge to a nursing home or to require 24-hour care.

Those patients assigned to usual care will receive written stroke preparedness education. This protocol will evaluate the effectiveness of this intervention to reduce blood pressure, and individual stroke risk factors and future stroke risk. Additionally, we will evaluate the ability of the these strategies to conduct education to affect positive change in taking medications as directed, stroke knowledge 6 months and 12 months after hospital admission, attendance at follow-up health care appointments, and cost-effectiveness. After 1 year participants will be followed quarterly for up to 3 years to track events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild ischemic cerebral infarction or mild intracerebral hemorrhage (NIHSS < 5) or TIA based on a clinical definition of focal neurologic deficits consistent with a single vascular territory of the brain
* Aged greater than 18 years at onset of event
* Resident of NY Metropolitan community in home with land or cell phone.
* Vascular risk factors including HTN history or elevated blood pressure (>130/85 mmHg) at the time of discharge, smoking, diabetes or metabolic syndrome
* Discharge to home
* English or Spanish Speaker

Exclusion Criteria:

* Patients unable to give informed consent
* Discharged to long-term nursing home or requiring 24 hour care.
* A Modified Rankin score > 2 at baseline
* Pre-stroke dementia history.
* Patients with end stage cancer, or other medical conditions resulting in mortality less than 1 year.
* Patient does not speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 6 months and 1 year
  change in overall blood pressure

SECONDARY OUTCOMES:
Secondary Incident | up to 3 years
  A secondary outcome is when the patient has a new visit to the ED or another hospital; admission that it is not a stroke/TIA nor ICH. Instead, it might be a seizure, headache, migraine, anything else neurological.

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Boden-Albala, DrPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - NYU Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082
- [Derived] Goldmann E, Jacoby R, Finfer E, Appleton N, Parikh NS, Roberts ET, Boden-Albala B. Positive Health Beliefs and Blood Pressure Reduction in the DESERVE Study. J Am Heart Assoc. 2020 May 5;9(9):e014782. doi: 10.1161/JAHA.119.014782. Epub 2020 Apr 28. PMID 32340524
- [Derived] Boden-Albala B, Goldmann E, Parikh NS, Carman H, Roberts ET, Lord AS, Torrico V, Appleton N, Birkemeier J, Parides M, Quarles L. Efficacy of a Discharge Educational Strategy vs Standard Discharge Care on Reduction of Vascular Risk in Patients With Stroke and Transient Ischemic Attack: The DESERVE Randomized Clinical Trial. JAMA Neurol. 2019 Jan 1;76(1):20-27. doi: 10.1001/jamaneurol.2018.2926. PMID 30304326